CLINICAL TRIAL: NCT03433924
Title: An Epidemiologic Study on PD-L1 Expression Combined With Clinical Observation of Initial Treatment Pattern and Overall Survival in the Chinese Muscle Invasive Urothelial Bladder Carcinoma Patients.
Brief Title: An Epidemiologic Study on PD-L1 Expression Combined With Clinical Observation in the Chinese MIUBC Patients.
Acronym: POLARIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9012R00001
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the study will collect sections for certain testing following the priority: PD-L1 (3 sections) > CD8 (2 sections) > TMB (6 sections). The minimal required sections number is 3, specially for PD-L1 testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Primary Objective of this observational study is to investigate the prevalence of high PD-L1 expression in Chinese MIUBC patients.

DETAILED DESCRIPTION:
The primary objective of this observational study is:

•To investigate the prevalence of high PD-L1 expression in Chinese MIUBC patients. High PD-L1 expression is defined as ≥25% tumor cell membrane positivity for PD-L1 at any intensity above background staining as noted on the corresponding negative control OR ≥25% tumor associated immune cell positivity for PD-L1 at any intensity above background staining as noted on the corresponding negative control.

Note: PD-L1 High (>=25% tumor cell membrane positivity for PD-L1 or 1) IF IC area >1%: >=25% tumor associated immune cell positivity for PD-L1; 2) If IC area=1%: 100% tumor associated immune cell positivity for PD-L1). PD-L1 Low if criteria not met for PD-L1 High.

The second objectives of this observational study are:

* To investigate the PD-L1 expression profile in TC or IC in Chinese MIUBC patients.
* To assess the concordance of PD-L1 testing results generated from the hospital labs with those from the central lab.
* To observe the initial treatment pattern for MIUBC patients in usual clinical practice in China.
* To observe 2-year OS of the Chinese MIUBC patients.

The exploratory objectives of this observational study are:

* To explore the relationship between the demographic characteristics and expression of PD-L1 and other exploratory biomarkers including immune cell (IC) subset CD8+ T cells and tumor mutation burden (TMB).
* To explore the relationship between OS and the demographic characteristics as well as the expression of biomarkers.
* To explore the relationship between PD-L1 and TMB, PD-L1 and CD8 positive T cell respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of screening.
* Be able and willing to sign the informed consent form (ICF).
* Patients with histologically or cytologically documented, muscle invasive urothelial carcinoma (ie, T2 toT4, any N, any M) of bladder (see National Comprehensive Cancer Network [NCCN] Bladder Cancer Guidelines), who had not been previously treated with any systemic chemotherapy, radiotherapy, investigational product, or biologic therapy for cancer treatment.
* For PD-L1 testing by IHC assay, all patients were able to provide a newly acquired tumor sample within 60 days before enrollment by cystectomy, transurethral resection or biopsy. Samples with limited tumor content and fine needle aspirate specimens were not acceptable. Specimens from metastatic bone lesions were typically unacceptable unless there was a significant soft tissue component. The tumor specimen submitted to establish PD-L1 status should be of sufficient quantity to allow for PD-L1 IHC analyses and was preferred in FFPE blocks.

Exclusion Criteria:

* Prior acquiring tumor tissue samples exposure to immune-mediated therapy (including Bacillus Calmette Guerin), including but not limited to, any anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti PD L2 antibodies, therapeutic anticancer vaccines.
* Any concurrent chemotherapy, investigational product, or biologic therapy for cancer treatment. Note: Local treatment of isolated lesions, excluding target lesions, for palliative intent was acceptable (eg, local surgery or radiotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of MIUBC
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
the prevalence of High PD-L1 expression in the MIUBC patients | Tumor tissue samples should be acquired within 60 days before the enrollment and available for testing.
  Tumor tissue will be collected from all eligible patients who sign the ICF. Samples will be tested for PD-L1 expression status.

SECONDARY OUTCOMES:
Proportion of patients with different PD-L1 expression level | Tumor tissue samples should be acquired within 60 days before the enrollment and available for testing.
  Proportion of patients with different PD-L1 expression level
PD-L1 testing concordance between central lab and hospital labs | Tumor tissue samples should be acquired within 60 days before the enrollment and available for testing.
  PD-L1 testing concordance between central lab and hospital labs
Distribution percent of different treatment approaches | enrollment visit
  Distribution percent of different treatment approaches
2-year OS | From enrollment to OS, up to 2 years
  follow up for OS up to 2 years from the baseline

OTHER OUTCOMES:
The prevalence of PD-L1 expression by subgroups | enrollment visit
  The prevalence of PD-L1 expression by subgroups according to age, gender, primary tumor site, metastatic disease, at baseline, and prior tobacco use, etc
OS by subgroups | from enrollment to OS, up to 2 years
  OS by subgroups according to age, gender, primary tumor site, metastatic disease at baseline and the PD-L1 expression of high and low/negative as well as other biomarkers, etc. Simple correlation coefficients among biomarkers including PD-L1 with TMB, PD-L1 with CD8+ T cell, PD-L1+ IC with CD8+ T cell.
Simple correlation coefficients among biomarkers | enrollment visit
  Simple correlation coefficients among biomarkers including PD-L1 with TMB, PD-L1 with CD8+ T cell, PD-L1 positive IC with CD8+ T cell.

CONTACTS AND LOCATIONS:
Overall Officials: Liqun ZHOU, doctor, Principal Investigator — Peking University First Hospital
Locations (14):
- China (14):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Meizhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: No
Chinese Laws and Regulations don't allow

REFERENCES:
- See also: CSR synopsis_redacted and confirmd by GSD — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9012R00001&attachmentIdentifier=620a24aa-cbcc-44e4-8581-76b171fa0b70&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=